CLINICAL TRIAL: NCT00515710
Title: A Long-Term Follow-Up Study in Subjects With Sever Hemophilia B Who Received Adeno-Associated Viral Vectors Expressing Human Factor IX
Brief Title: LTFU for Gene Transfer Subjects With Hemophilia B
Status: Completed | Type: Observational
Sponsor: Spark Therapeutics, Inc. (Industry)
Collaborators: Children's Hospital of Philadelphia (Other); The Hemophilia Center of Western Pennsylvania (Other); Royal Prince Alfred Hospital, Sydney, Australia (Other)
Responsible Party: Sponsor
Other Study IDs: AAV2-hFIX16-LTFU-01
Record Dates: First submitted 2007-08-10; First posted 2007-08-14 (Estimated); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Hemophilia B
Keywords: Hemophilia B; Gene Transfer; Adeno-Associated Virus (AAV); Coagulation Factor IX; Long-term Follow-up; Delayed Adverse Events
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Prior gene therapy study subjects receiving AAV2-hFIX16.

SUMMARY:
Several subjects enrolled in a multi-site, gene transfer clinical study to evaluate the intrahepatic administration of AAV2-hFIX16 vector for the treatment of severe hemophilia B between 2001 and 2009. As the US FDA has established guidelines for the long-term follow-up (LTFU) of subjects receiving investigational gene therapy products, this protocol seeks to characterize the clinical outcome and the type and seriousness of adverse events following the AAV gene transfer. The primary study tools will consist of annual history/physical examination and blood tests, as well as periodic liver ultrasound, to characterize clinical outcomes. Where possible, data will be obtained for up to 15 years following hepatic AAV2-hFIX16 gene transfer.

DETAILED DESCRIPTION:
A prior clinical gene transfer study of intrahepatic adeno-associated virus (AAV) vector administration of the factor IX gene (AAV2-hFIX16) to adult subjects with severe hemophilia B enrolled several subjects from 2001 through 2004. These subjects received various doses of AAV2-hFIX16 manufactured by Avigen, Inc. (Alameda, CA). They were monitored up to at least one year following vector administration for evaluation of adverse events and for indices of efficacy. At the time study enrollment was suspended by Avigen, Inc., and IND 9398 under which the study was conducted was transferred to The Children's Hospital of Philadelphia (May 2005), there were no guidelines for long-term follow-up of the trial subjects. However, in an unrelated study conducted in France, of pediatric subjects administered integrating retrovirus vectors for X-linked severe combined immune deficiency (X-SCID), several leukemias developed years after transfer of the γc common chain gene. The underlying mechanism was attributed to proviral integration near, and upregulation of, proto-oncogenes such as LMO-2, coupled with robust expression of the γc common chain, inducing unregulated cellular proliferation. In response to these events, and in concert with the NIH and gene transfer scientific community, the U.S. Food and Drug Administration (US FDA) issued guidelines for the 'long-term follow-up of gene transfer subjects'. Since AAV vectors have a low rate of genomic integration, the risks of integration are low, but the long-term effect of the persistence of vector particles in humans is unknown. The investigators plan to enroll available subjects from the prior intrahepatic AAV gene transfer study to this observational study to follow them for up to 15 years after gene transfer.

An additional subject received AAV2-hFIX16 vector, manufactured by CCMT at CHOP, via hepatic artery infusion in January 2009. The study AAV2-hFIX-002, an amendment to the prior Avigen, Inc. clinical protocol modified to include transient immunomodulation, was conducted under IND 9398. This subject was monitored for three years following vector administration under clinical study AAV2-hFIX-002; amendment one of the current protocol transfers his annual long-term follow-up visits to AAV2-hFIX16-LTFU-01.

Spark Therapeutics will be the study sponsor; prior vector administration sites or referral/follow up sites will participate as study sites. The long-term follow-up (LTFU) study will consist primarily of endpoints including annual history, physical examination, blood tests, urinalysis, and periodic liver ultrasound. Adverse event reporting will focus on the development of oncologic, hematologic, neurologic and auto-immune events following gene transfer as specified in the November 2006 FDA Center for Biologics Evaluation and Research (CBER) guidance document entitled, "Gene Therapy Clinical Trials - Observing Subjects for Delayed Adverse Events."1 The LTFU study seeks to provide longitudinal information, and should adverse events occur, more timely discovery and treatment.

ELIGIBILITY:
Inclusion Criteria

-Adult subjects who participated in prior intrahepatic AAV2-hFIX16 gene transfer studies

Exclusion Criteria

* Subjects who will not consent for study
* Subjects who the investigators believe are not capable of performing endpoints of the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prior gene therapy study subjects receiving AAV2-hFIX16.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2007-08; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of intra-hepatic administration of AAV2-hFIX. Toxicity related to the administration of AAV2-hFIX will be evaluated locally and systemically. | Long-term follow-up up to 15 years
  Annual study visits will be comprised of history, physical examination, blood tests and urinalysis and may include hepatic ultrasound tests; additional medical information may be needed to determine the relationship of adverse events to the investigational gene therapy vector AAV2-hFIX16.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Director, Study Director — Spark Therapeutics, Inc.
Locations (2):
- United States (2):
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Hemophilia Center of Western Pennsylvania, Pittsburgh, Pennsylvania